CLINICAL TRIAL: NCT04061317
Title: A Pilot Study to exPlOre the exisTence and Impact of FRAILTY in Patients Over the Age of 70 Undergoing Cardiac Interventions
Brief Title: SPOT-FRAILTY Assessment of Frailty in Patients Over the Age of 70 Undergoing a Cardiac Intervention
Acronym: SPOT FRAILTY
Status: Terminated | Type: Observational
Why Stopped: COVID Restrictions in a vulnerable population.
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Burdett Trust for Nursing (Other)
Responsible Party: Sponsor
Other Study IDs: V1 - 08-04-2019
Record Dates: First submitted 2019-04-15; First posted 2019-08-19 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Frailty Assessment — We will use validated measures to determine existence of frailty prior to interventional cardiac procedures (PRISMA-7, Edmonton and FRIED Frailty Index). We will repeat the measures at 6 weeks and 6 months post procedure. We will also collect clinical data to assess any links between frailty and clinical outcomes.
  We are also keen to understand the effects of health-related quality of life on frailty and will be collecting generic data via the SF-36 and EQ5-D.
  Other Names: Quality of Life Assessment

SUMMARY:
Rocha (2017), published a systematic review and meta-analysis highlighting the clinical utility of frailty scales for the prediction of post-operative complications. The results of the review of 15 studies show that, overall, frailty significantly increases the risk for developing adverse outcomes such as, mortality, morbidity and extended length of hospital stay. However, different frailty scales showed different prevalence of frailty even when tested in the same population, which means that future studies are required for a better understanding of frailty tools. Early detection of frailty may provide a window of opportunity for intervention and a key factor to determine clinical outcomes.

DETAILED DESCRIPTION:
The investigators anticipate that this project will allow the creation of a registry to describe our population in terms of the presence or absence of frailty. The investigators will use validated measures to determine existence of frailty prior to interventional cardiac procedures (PRISMA-7, Edmonton and FRIED Frailty Index). The measures will be repeated at 6 weeks and 6 months post procedure. Clinical data will also be collected to assess any links between frailty and clinical outcomes. Data collection sheets will be designed, data will be entered and analyzed by a statistician.. If the data provides meaningful insight, the investigator will aim to create a specific frailty tool for the cardiac population.

The investigators are also keen to understand the effects of health-related quality of life on frailty and will be collecting generic data via the SF-36 and EQ5-D. In order to assess the lived experience of frailty, the investigators are proposing a qualitative interview for 15 willing patients, to allow the exploration of the concepts of frailty in more detail for patients who have undergone a cardiac intervention.

The totality of the data collection will help the study team examine care pathways and assess any areas of concern, which may be addressed for the benefit of patients in the future.

Once we have gathered data to define the population in terms of frailty and the impact of frailty on health-related quality of life, the investigators aim to adapt the services to accommodate the needs of frail patients undergoing heart procedures. This may involve amended pre-admission care which may influence discharge planning, depending on the nature of the individual patients. An integrated care pathway (ICP) is a step by step approach to patient care which also considers the requirements of research, training, resources, clinical governance and performance. It is anticipated that an amended ICP may be created for patients with frailty. . This initial project will form part of a longer-term plan to assess and manage frailty in a systematic process.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 70 and above
2. Scheduled to receive an elective cardiac procedure.
3. Willing to undergo frailty assessment
4. Able to walk with or without aids.
5. Willingness to attend a 6 week and 6 months follow up appointments.
6. Able to provide full informed consent. -

Exclusion Criteria:

1. Unable to provide informed consent
2. Scheduled to receive an emergency procedure -

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients aged 70 years and above scheduled to receive an elective cardiac intervention.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of frailty in a population undergoing cardiac intervention | Baseline, 6 weeks and 6 months post procedure
  The primary endpoint is to describe our population related to validated frailty assessment tools and explore any associations with a generic quality of life measure.
  As above

SECONDARY OUTCOMES:
Frailty assessment via the FRIED criteria | Baseline, 6 weeks and 6 months post procedure
  Assessment using the FRIED frailty tool
Frailty assessment via the EDMONTON frailty criteria | Baseline, 6 weeks and 6 months post procedure
  Assessment using the EDMONTON frailty criteria
Frailty assessment via the PRISMA frailty score | Baseline, 6 weeks and 6 months post procedure
  Assessment using the PRISMA frailty tool

CONTACTS AND LOCATIONS:
Overall Officials: Paula Rogers, RGN, BSc, MSc, Principal Investigator — Royal Brompton and Harefield NHS Foundation Trust
Locations (1):
- Harefield Hospital, Harefield, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided